CLINICAL TRIAL: NCT02807636
Title: A Phase III, Multicenter, Randomized, Placebo-Controlled Study of Atezolizumab (Anti-PD-L1 Antibody) as Monotherapy and in Combination With Platinum-Based Chemotherapy in Patients With Untreated Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: Study of Atezolizumab as Monotherapy and in Combination With Platinum-Based Chemotherapy in Participants With Untreated Locally Advanced or Metastatic Urothelial Carcinoma
Acronym: IMvigor130
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WO30070; 2016-000250-35 (EudraCT Number)
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Results first posted 2023-12-13 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial carcinoma; Bladder cancer; Anti-PD-L1; Transitional carcinoma; Tecentriq; Atezolizumab; IMvigor130
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — atezolizumab; Carboplatin; Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Atezolizumab+Gemcitabine+Carboplatin/Cisplatin (Experimental): Participants will receive blinded atezolizumab in combination with open-label platinum-based chemotherapy (gemcitabine with either cisplatin or carboplatin).
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Gemcitabine; Drug: Cisplatin
- Placebo+Gemcitabine+Carboplatin/Cisplatin (Placebo Comparator): Participants will receive blinded placebo matched to atezolizumab in combination with open-label platinum-based chemotherapy (gemcitabine with either cisplatin or carboplatin).
  Interventions: Drug: Carboplatin; Drug: Gemcitabine; Other: Placebo; Drug: Cisplatin
- Atezolizumab Monotherapy (Experimental): Eligible participants will receive open-label atezolizumab as monotherapy.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a fixed dose of 1200 milligrams (mg) by intravenous (IV) infusion on Day 1 of each 21-day cycle until investigator-assessed disease progression per RECIST v1.1. In specific circumstances treatment may continue beyond disease progression.
  Other Names: Tecentriq
  Arms: Atezolizumab Monotherapy; Atezolizumab+Gemcitabine+Carboplatin/Cisplatin
Drug: Carboplatin — Carboplatin will be administered at doses to achieve area under the concentration-time curve (AUC) of 4.5 milligram per milliliter into minute (mg/mL*min) by IV infusion on Day 1 of each 21-day cycle until investigator-assessed disease progression per RECIST v1.1 or unacceptable toxicity.
  Arms: Atezolizumab+Gemcitabine+Carboplatin/Cisplatin; Placebo+Gemcitabine+Carboplatin/Cisplatin
Drug: Gemcitabine — Gemcitabine will be administered at a dose of 1000 milligrams per square meter (mg/m^2) by IV infusion on Day 1 and Day 8 of each 21-day cycle, until investigator-assessed disease progression per RECIST v1.1 or unacceptable toxicity.
  Arms: Atezolizumab+Gemcitabine+Carboplatin/Cisplatin; Placebo+Gemcitabine+Carboplatin/Cisplatin
Other: Placebo — Placebo matched to atezolizumab will be administered by IV infusion on Day 1 of each 21-day cycle until investigator-assessed disease progression per RECIST v1.1. In specific circumstances treatment may continue beyond disease progression.
  Arms: Placebo+Gemcitabine+Carboplatin/Cisplatin
Drug: Cisplatin — Cisplatin will be administered at a dose of 70 mg/m^2 by IV infusion on Day 1 of each 21-day cycle until investigator-assessed disease progression per RECIST v1.1 or unacceptable toxicity.
  Arms: Atezolizumab+Gemcitabine+Carboplatin/Cisplatin; Placebo+Gemcitabine+Carboplatin/Cisplatin

SUMMARY:
A Phase III, randomised study of atezolizumab alone and in combination with chemotherapy versus chemotherapy alone in participants with untreated advanced urothelial cancer.

ELIGIBILITY:
Inclusion Criteria

* Considered to be eligible to receive platinum-based chemotherapy, in the investigator's judgment
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to (</=) 2
* Histologically documented, locally advanced (T4b, any N; or any T, N2-3) or metastatic urothelial carcinoma (mUC) (M1, Stage IV) (also termed transitional cell carcinoma [TCC] or urothelial cell carcinoma [UCC] of the urinary tract; including renal pelvis, ureters, urinary bladder, and urethra)
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (blocks preferred) or at least 15 unstained slides, with an associated pathology report, for central testing and determined to be evaluable for tumor PD-L1 expression prior to study enrollment; participants who have fewer than 15 unstained slides available at baseline (but no less than [<] 10) may be eligible following discussion with the Medical Monitor
* No prior chemotherapy for inoperable locally advanced or mUC
* For participants who received prior adjuvant/neoadjuvant chemotherapy or chemo-radiation for urothelial carcinoma, a treatment-free interval more than (>) 12 months between the last treatment administration and the date of recurrence is required in order to be considered treatment naive in the metastatic setting
* Prior local intravesical chemotherapy or immunotherapy is allowed if completed at least 4 weeks prior to the initiation of study treatment
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 6 months after the last dose of carboplatin, cisplatin, or gemcitabine or for 5 months after the last dose of atezolizumab
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm

Exclusion Criteria:

* Any approved anti-cancer therapy, including chemotherapy or hormonal therapy, within 3 weeks prior to initiation of study treatment
* Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 28 days prior to enrolment
* Active or untreated CNS metastases as determined by computed tomography (CT) or magnetic resonance imaging evaluation during screening and prior radiographic assessments
* Participants with treated asymptomatic central nervous system (CNS) metastases are eligible, provided they meet all of the following criteria: * Evaluable or measurable disease outside the CNS * No metastases to midbrain, pons, medulla, or within 10 mm of the optic apparatus (optic nerves and chiasm) * No history of intracranial or spinal cord hemorrhage * No ongoing requirement for corticosteroid as therapy for CNS disease; anti-convulsants at a stable dose are allowed * No evidence of significant vasogenic edema * No stereotactic radiation, whole-brain radiation or neurosurgical resection within 4 weeks prior to Cycle 1, Day 1 * Radiographic demonstration of interim stability (i.e., no progression) between the completion of CNS-directed therapy and the screening radiographic study * Screening CNS radiographic study >/=4 weeks since completion of radiotherapy or surgical resection and >/=2 weeks since discontinuation of corticosteroids
* Prior treatment with CD137 agonists, anti-CTLA-4, anti-programmed death-1 (PD-1), or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1, Day 1 or anticipated requirement for systemic immunosuppressive medications during the study
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Uncontrolled tumour-related pain or hypercalcemia
* Significant cardiovascular disease including known left ventricular ejection fraction (LVEF) <40%
* Severe infections within 4 weeks before randomization or therapeutic oral or IV antibiotics within 2 weeks before randomization
* Major surgical procedure within 4 weeks prior to randomization or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis
* Malignancies other than urothelial carcinoma within 5 years prior to Cycle 1, Day 1
* Life expectancy of <12 weeks
* Pregnant or lactating, or intending to become pregnant during the study
* Serum albumin <25 gram per liter (g/L)
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease
* Participants with prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan
* Positive test for human immunodeficiency virus (HIV)
* Active hepatitis B or hepatitis C
* Active tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1213 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (204):
- United States (18):
  - Highlands Oncology Group, Rogers, Arkansas
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Yale School of Medicine, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Christina Care Institutional Review Board, Newark, Delaware
  - Florida Cancer Specialists, Fort Myers, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Florida Cancer Specialists (St. Petersburg ? St. Anthony?s Professional Building), St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Parkview Research Center, Fort Wayne, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - East Jefferson Hematology Oncology, Metairie, Louisiana
  - Park Nicollet Clin-Cancer Ctr, Saint Louis Park, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Mount Sinai School of Medicine - Tisch Cancer Institute, New York, New York
  - University of North Carolina, Lineberger Cancer Ctr, Chapel Hill, North Carolina
  - Bon Secours - St. Francis Hospital, Greenville, South Carolina
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
- Australia (6):
  - Macquarie University Hospital, Macquarie University, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Lyell McEwin Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Cabrini Medical Centre, Malvern, Victoria
  - Sunshine Hospital, St Albans, Victoria
- Belgium (4):
  - GHdC Site Notre Dame, Charleroi
  - AZ Sint Lucas (Sint Lucas), Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - CHC MontLégia, Liège
- Clinical center University of Sarajevo, Sarajevo, Bosnia and Herzegovina
- Brazil (11):
  - CETUS Hospital Dia Oncologia, Belo Horizonte, Minas Gerais
  - Hospital Luxemburgo, Belo Horizonte, Minas Gerais
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Clinica Viver, Santa Maria, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Beneficencia Portuguesa de Sao Paulo, São Paulo, São Paulo
  - Clinicas Oncologicas Integradas - COI, Rio de Janeiro
- Canada (7):
  - Arthur J.E. Child Comprehensive Cancer Center-Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, CSI, Kelowna, British Columbia
  - Dr. Georges L. Dumont University Hospital Centre, Moncton, New Brunswick
  - Juravinski Cancer Clinic, Hamilton, Ontario
  - Lakeridge Health Center, Oshawa, Ontario
  - North York General Hospital, Toronto, Ontario
- Chile (4):
  - Bradford Hill Centro de Investigaciones Clinicas, Recoleta
  - OrlandiOncología, Santiago
  - Fundacion Arturo Lopez Perez, Santiago
  - Clinica Alemana, Vitacura
- China (9):
  - Beijing Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Chongqing Cancer Hospital, Chongqing
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - The 2nd Hospital of Tianjin Medical University, Tianjin
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
  - University Hospital Motol, Prague
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
- Finland (2):
  - Oulu University Hospital, Oulu
  - Turku Uni Central Hospital, Turku
- Georgia (2):
  - Research institute for Clinical Medicine, Tbilisi
  - National Center of Urology, Tbilisi
- Greece (2):
  - Alexandras General Hospital of Athens, Athens
  - University Hospital of Patras Medical Oncology, Pátrai
- Hong Kong (4):
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - The Chinese University of Hong Kong, Hong Kong
- Rambam Health Care Campus, Haifa, Israel
- Italy (12):
  - IRCCS Ospedale Casa Sollievo Della Sofferenza, San Giovanni Rotondo, Apulia
  - Azienda Ospedaliera A. Cardarelli, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena, Modena, Emilia-Romagna
  - Policlinico Umberto i di Roma, Rome, Lazio
  - Az. Osp. Uni Ria San Martino, Genoa, Liguria
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - A.O CITTA' DELLA SALUTE E DELLA SCIENZA D. - Presidio San Lazzaro, Turin, Piedmont
  - Azienda USL8 Arezzo-Presidio Ospedaliero 1 San Donato, Arezzo, Tuscany
  - Azienda Ospedaliera S. Maria - Terni, Terni, Umbria
  - IRCCS Istituto Oncologico Veneto (IOV), Padua, Veneto
- Japan (14):
  - Nagoya University Hospital, Aichi
  - Hirosaki University Hospital, Aomori
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - Gunma University Hospital, Gunma
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - University of Tsukuba Hospital, Ibaraki
  - Kanazawa University Hospital, Ishikawa
  - Kumamoto University Hospital, Kumamoto
  - Niigata University Medical & Dental Hospital, Niigata
  - Osaka Metropolitan University Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Toranomon Hospital, Tokyo
  - The Cancer Institute Hospital, JFCR, Tokyo
  - Keio University Hospital, Tokyo
- Malaysia (2):
  - Hospital Kuala Lumpur, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur, FED. Territory of Kuala Lumpur
- Mexico (4):
  - Consultorio Médico, Zapopan, Jalisco
  - Health Pharma Professional Research, CD Mexico, Mexico CITY (federal District)
  - IMSS Hospital General de Zona No. 48 S. Pedro Xalpa, Mexico CITY (federal District), Mexico CITY (federal District)
  - Cancerología, Querétaro
- Netherlands (4):
  - Martini Ziekenhuis, Groningen
  - Hagaziekenhuis, locatie Leyweg, NL -DEN HAAG
  - Zuyderland Medisch Centrum, Sittard-Geleen
  - Isala Klinieken, Sophia, Zwolle
- Poland (7):
  - Bialostockie Centrum Onkologii, Bialystok
  - Przychodnia Lekarska KOMED, Roman Karaszewski, Konin
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Woj.Wielospecjalistyczne Centrum Onkologii i Traumatologii, Lodz
  - Oddzial Chemioterapii Szpitala Klinicznego Nr 1 w Poznaniu, Poznan
  - NU-MED Centrum Diagnostyki i Terapii Onkologicznej, Tomaszów Mazowiecki
  - Szpital Grochowski im. dr med. Rafa?a Masztaka Sp. z o.o., Warsaw
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - IPO do Porto, Porto
- Romania (3):
  - Spitalul Judetean de Urgenta Dr Constantin Opris, Baia Mare
  - Institute Of Oncology Bucharest, Bucharest
  - Oncology Center Sf. Nectarie, Craiova
- Russia (9):
  - SBEI of HPE ?Bashkir State Medical University? of MoH RF, Ufa, Bashkortostan Republic
  - Krasnoyarsk Regional Oncology Dispensary n.a. Krizhanovsky, Krasnoyarsk, Krasnodarskiy Kray
  - Blokhin Cancer Research Center, Moscow, Moscow Oblast
  - Russian Scientific Center of Roentgenoradiology, Moscow, Moscow Oblast
  - P.A. Herzen Oncological Inst., Moscow, Moscow Oblast
  - Privolzhsk Regional Medical Center, Nizhny Novgorod, Niznij Novgorod
  - SBEI HPE "The First St.Petersburg State Medical University n.a. acad. I.P.Pavlova"of MoH of RF, Saint Petersburg, Sankt-Peterburg
  - Sverdlovsk Regional Clinical Hospital 1, Yekaterinburg, Sverdlovsk Oblast
  - Ivanovo Regional Oncology Dispensary, Ivanovo
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
  - Clinical Centre Nis, Clinic for Oncology, Niš
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
  - Oncocare Cancer Centre, Singapore
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Africa (3):
  - Cancercare, Port Elizabeth
  - Wilgers Oncology Centre, Pretoria
  - Sandton Oncology Medical Group, Sandton
- South Korea (4):
  - Kyungpook National University Medical Center, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (32):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Complejo Hospitalario de Althaia, Manresa, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Provincial de Castellon, Castellon, Castellon
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital de Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clinic de Barcelona. Unidad de Nuevas Terapias, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institutio Catalan De Oncologia, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Complejo Asistencial Universitario De Burgos, Burgos
  - Hospital San Pedro De Alcantara, Cáceres
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico, Jaén
  - Complejo Asistencial Universitario de Leon, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario de Toledo, Toledo
  - Hospital Universitario la Fe, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (6):
  - Chang Gung Medical Foundation - Kaohsiung, Kaohisung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung Uni Hospital, Tainan
  - National Taiwan Uni Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou, Urinary Oncology, Taoyuan District
- Thailand (4):
  - Vajira Hospital, Bangkok
  - Chulalongkorn Hospital, Bangkok
  - Faculty of Med. Siriraj Hosp., Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- Turkey (Türkiye) (7):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital, Adana
  - Ankara Bilkent City Hospital, Ankara
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Bezmi Alem Vakif University Medical School, Istanbul
  - Istanbul University Cerrahpa?a-Cerrahpa?a Medical Faculty, Istanbul
  - Hacettepe Uni Medical Faculty Hospital, S?hhiye, Ankara
  - 19 Mayis University Medical Faculty, Samsun
- Ukraine (3):
  - Regional Clinical Center of Urology and Nephrology n.a. V.I. Shapoval Department of Urology #4, Kharkiv, Kharkiv Governorate
  - CI Dnipropetrovsk CMCH #4 MA of MOHU Ch of Oncology and MR, Dnipropetrovsk
  - Zaporizhzhia Regional Clinic, Zaporizhzhia
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - The York Hospital, York

REFERENCES:
- [Derived] Galsky MD, Guan X, Rishipathak D, Rapaport AS, Shehata HM, Banchereau R, Yuen K, Varfolomeev E, Hu R, Han CJ, Li H, Liang Y, Vucic D, Wang L, Zhu J, Yu H, Herbst RH, Hajaj E, Kiner E, Bamias A, De Santis M, Davis ID, Arranz JA, Kikuchi E, Bernhard S, Williams P, Lee C, Mellman I, Sanjabi S, Johnston R, Black PC, Grande E, Mariathasan S. Immunomodulatory effects and improved outcomes with cisplatin- versus carboplatin-based chemotherapy plus atezolizumab in urothelial cancer. Cell Rep Med. 2024 Feb 20;5(2):101393. doi: 10.1016/j.xcrm.2024.101393. Epub 2024 Jan 26. PMID 38280376
- [Derived] Grande E, Arranz JA, De Santis M, Bamias A, Kikuchi E, Del Muro XG, Park SH, De Giorgi U, Alekseev B, Mencinger M, Izumi K, Schutz FA, Puente J, Li JR, O'Donnell PH, Kalebasty AR, Ye D, Mariathasan S, Bene-Tchaleu F, Bernhard S, Lee C, Davis ID, Galsky MD. Atezolizumab plus chemotherapy versus placebo plus chemotherapy in untreated locally advanced or metastatic urothelial carcinoma (IMvigor130): final overall survival analysis results from a randomised, controlled, phase 3 study. Lancet Oncol. 2024 Jan;25(1):29-45. doi: 10.1016/S1470-2045(23)00540-5. Epub 2023 Dec 12. PMID 38101433
- [Derived] Bamias A, Davis ID, Galsky MD, Arranz JA, Kikuchi E, Grande E, Del Muro XG, Park SH, De Giorgi U, Alekseev B, Mencinger M, Izumi K, Schutz FA, Puente J, Li JR, Panni S, Gumus M, Ozguroglu M, Mariathasan S, Poloz Y, Bene-Tchaleu F, Lee C, Bernhard S, De Santis M. Atezolizumab monotherapy versus chemotherapy in untreated locally advanced or metastatic urothelial carcinoma (IMvigor130): final overall survival analysis from a randomised, controlled, phase 3 study. Lancet Oncol. 2024 Jan;25(1):46-61. doi: 10.1016/S1470-2045(23)00539-9. Epub 2023 Dec 12. PMID 38101431
- [Derived] Grande E, Bamias A, Galsky MD, Kikuchi E, Davis ID, Arranz JA, Rezazadeh Kalebasty A, Garcia Del Muro X, Park SH, De Giorgi U, Alekseev B, Mencinger M, Izumi K, Puente J, Li JR, Bernhard S, Nicholas A, Telliez J, De Santis M. Overall Survival by Response to First-line Induction Treatment with Atezolizumab plus Platinum-based Chemotherapy or Placebo plus Platinum-based Chemotherapy for Metastatic Urothelial Carcinoma. Eur Urol Open Sci. 2023 Nov 4;58:28-36. doi: 10.1016/j.euros.2023.10.002. eCollection 2023 Dec. PMID 37954037
- [Derived] Galsky MD, Arija JAA, Bamias A, Davis ID, De Santis M, Kikuchi E, Garcia-Del-Muro X, De Giorgi U, Mencinger M, Izumi K, Panni S, Gumus M, Ozguroglu M, Kalebasty AR, Park SH, Alekseev B, Schutz FA, Li JR, Ye D, Vogelzang NJ, Bernhard S, Tayama D, Mariathasan S, Mecke A, Thastrom A, Grande E; IMvigor130 Study Group. Atezolizumab with or without chemotherapy in metastatic urothelial cancer (IMvigor130): a multicentre, randomised, placebo-controlled phase 3 trial. Lancet. 2020 May 16;395(10236):1547-1557. doi: 10.1016/S0140-6736(20)30230-0. PMID 32416780
- [Derived] Balar AV, Galsky MD, Rosenberg JE, Powles T, Petrylak DP, Bellmunt J, Loriot Y, Necchi A, Hoffman-Censits J, Perez-Gracia JL, Dawson NA, van der Heijden MS, Dreicer R, Srinivas S, Retz MM, Joseph RW, Drakaki A, Vaishampayan UN, Sridhar SS, Quinn DI, Duran I, Shaffer DR, Eigl BJ, Grivas PD, Yu EY, Li S, Kadel EE 3rd, Boyd Z, Bourgon R, Hegde PS, Mariathasan S, Thastrom A, Abidoye OO, Fine GD, Bajorin DF; IMvigor210 Study Group. Atezolizumab as first-line treatment in cisplatin-ineligible patients with locally advanced and metastatic urothelial carcinoma: a single-arm, multicentre, phase 2 trial. Lancet. 2017 Jan 7;389(10064):67-76. doi: 10.1016/S0140-6736(16)32455-2. Epub 2016 Dec 8. PMID 27939400

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 221 sites in 35 countries.
Pre-assignment Details: Stage 1 included atezolizumab+gemcitabine+carboplatin arm or placebo+gemcitabine+carboplatin arm. Participants ineligible for cisplatin-based chemo were enrolled in this stage. Stage 2 included addition of atezolizumab monotherapy arm and allowed participants who were eligible for cisplatin-based chemotherapy. Study is considered "Completed" because all pre-planned study analyses have been preformed for primary and secondary endpoints.
Groups:
- Placebo+Gemcitabine+Carboplatin/Cisplatin: Participants received blinded placebo matched to atezolizumab in combination with open-label platinum-based chemotherapy (gemcitabine with either cisplatin or carboplatin).
- Atezolizumab+Gemcitabine+Carboplatin/Cisplatin: Participants received blinded atezolizumab in combination with open-label platinum-based chemotherapy (gemcitabine with either cisplatin or carboplatin).
- Atezolizumab Monotherapy: Eligible participants received open-label atezolizumab as monotherapy.
Period: Overall Study
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Started | 400 | 451 | 362
Completed | 0 | 0 | 0
Not Completed | 400 | 451 | 362
Not completed — Lost to Follow-up | 10 | 13 | 6
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Symptomatic Deterioration | 0 | 1 | 0
Not completed — Withdrawal by Subject | 39 | 28 | 24
Not completed — Death | 303 | 332 | 272
Not completed — Study Terminated By Sponsor | 47 | 76 | 60
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy | Total
Number analyzed (Participants) | 400 | 451 | 362 | 1213
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.4 (9.5) | 67.5 (9.7) | 67.0 (9.1) | 67.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 113 | 82 | 297
  Male | 298 | 338 | 280 | 916
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 41 | 40 | 125
  Not Hispanic or Latino | 350 | 402 | 311 | 1063
  Unknown or Not Reported | 6 | 8 | 11 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 2 | 9
  Asian | 85 | 90 | 94 | 269
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 6 | 1 | 7
  White | 305 | 346 | 260 | 911
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 7 | 5 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Investigator Assessed Progression-Free Survival (PFS) in the Placebo+Gemcitabine+Carboplatin/Cisplatin Arm Versus Atezolizumab +Gemcitabine+Carboplatin/Cisplatin Arm
Description: PFS is defined as the time from randomization to the first documented disease progression as determined by the investigator with the use of RECIST v1.1, or death from any cause, whichever occurs first.
Time Frame: Baseline up to first documented disease progression or death, whichever occurs first (up to approximately 35 months)
Population: The ITT population was defined as all participants randomized to the Atezolizumab+Gemcitabine+Carboplatin/Cisplatin arm or the Placebo+Gemcitabine+Carboplatin/Cisplatin arm in Stages 1 and 2, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin
Number analyzed (Participants) | 400 | 451
Months | 6.34 [6.24 to 7.00] | 8.18 [6.51 to 8.34]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab+Gemcitabine+Carboplatin/Cisplatin; Stratification factors: Enrollment stage, PD-L1 status, Bajorin risk score/presence of liver metastases, and investigator choice of chemotherapy; Test type: Superiority; p = 0.0073, Log Rank — inverse normal combination; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.70 to 0.96]

2. Primary Outcome: Overall Survival (OS) in Atezolizumab+Gemcitabine+Carboplatin/Cisplatin Arm Versus Placebo+Gemcitabine+Carboplatin/Cisplatin Arm
Description: OS is defined as the time from randomization to death due to any cause.
Time Frame: Baseline until death due to any cause (up to approximately 73 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin
Number analyzed (Participants) | 400 | 451
Months | 13.44 [11.99 to 15.34] | 16.13 [14.19 to 18.76]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab+Gemcitabine+Carboplatin/Cisplatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0230, Regression, Cox — one-sided, inverse normal combination; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.73 to 1.0]

3. Primary Outcome: Overall Survival (OS) in Atezolizumab Monotherapy Arm Versus Placebo+Gemcitabine+Carboplatin/Cisplatin Arm
Description: OS is defined as the time from randomization to death due to any cause.
Time Frame: Baseline until death due to any cause (up to approximately 73 months)
Population: The ITT population includes only participants concurrently enrolled in Stage 2 and only those who had been randomized at the time of approval of Protocol WO30070 v6.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 359 | 360
Months | 13.34 [11.89 to 15.61] | 15.21 [13.14 to 17.68]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab Monotherapy; Stratification factors: PD-L1 status, Bajorin risk score/presence of liver metastases, and investigator choice of chemotherapy; Test type: Superiority; p = 0.3968, Log Rank; one-sided; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.82 to 1.16]

4. Secondary Outcome: Objective Response Rate (ORR) in Atezolizumab+Gemcitabine+Carboplatin/Cisplatin Arm Versus Placebo+Gemcitabine+Carboplatin/Cisplatin Arm
Description: Objective response rate (ORR) is defined as the proportion of participants with a confirmed objective response, either complete response (CR) or partial response (PR), observed on two assessments >= 28 days apart per RECIST v1.1, based on investigator assessment. The analysis population for ORR will be all randomized participants with measurable disease at baseline.
Time Frame: Baseline up to disease progression, death, or loss of follow-up, whichever occurs first (up to approximately 73 months)
Population: The ITT population was defined as all participants randomized to the Atezolizumab+Gemcitabine+Carboplatin/Cisplatin arm or the Placebo+Gemcitabine+Carboplatin/Cisplatin arm in Stages 1 and 2, whether or not the assigned study treatment was received. The measurable disease populations were defined as participants in the respective ITT populations with at least one measurable lesion according to RECIST v1.1 based on investigator assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin
Number analyzed (Participants) | 397 | 447
Percentage of Participants | 44.8 [39.87 to 49.88] | 48.1 [43.38 to 52.84]

5. Secondary Outcome: Objective Response Rate (ORR) in Atezolizumab Monotherapy Arm Versus Placebo+Gemcitabine+Carboplatin/Cisplatin Arm
Description: as for outcome 4
Time Frame: Baseline up to disease progression, death, or loss of follow-up, whichever occurs first (up to approximately 73 months)
Population: The ITT population includes only participants concurrently enrolled in Stage 2 and only those who had been randomized at the time of approval of Protocol WO30070 v6. The measurable disease populations were defined as participants in the respective ITT populations with at least one measurable lesion according to RECIST v1.1 based on investigator assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 356 | 359
Percentage of Participants | 44.4 [39.15 to 49.71] | 24.2 [19.89 to 29.01]

6. Secondary Outcome: Duration of Response (DOR) in Atezolizumab+Gemcitabine+Carboplatin/Cisplatin Arm Versus Placebo+Gemcitabine+Carboplatin/Cisplatin Arm
Description: Duration of response (DOR) is defined for participants with an objective response as the time from the first documented objective response to documented disease progression per RECIST v1.1, based on investigator assessment, or death due to any cause, whichever occurs first.
Time Frame: From first documented objective response (CR or PR) to disease progression, death, or loss of follow-up, whichever occurs first (up to approximately 73 months)
Population: The duration of response (DOR)-evaluable population is defined as participants with an objective response in the Atezolizumab+Gemcitabine+Carboplatin/Cisplatin arm or the Placebo+Gemcitabine+Carboplatin/Cisplatin arm in Stages 1 and 2.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin
Number analyzed (Participants) | 178 | 215
Months | 8.15 [6.34 to 8.61] | 9.13 [8.02 to 10.64]

7. Secondary Outcome: Duration of Response (DOR) in Atezolizumab Monotherapy Arm Versus Placebo+Gemcitabine+Carboplatin/Cisplatin Arm
Description: as for outcome 6
Time Frame: as for outcome 6
Population: The duration of response (DOR)-evaluable population is defined as participants with an objective response in the the ITT population which included only participants concurrently enrolled in Stage 2 and only those who had been randomized at the time of approval of Protocol WO30070 v6.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 158 | 87
Months | 8.11 [6.28 to 8.54] | 29.63 [15.90 to NA] — Upper CI limit is not evaluable because there were not enough events at later time to get a reliable upper CI.

8. Secondary Outcome: IRF-PFS
Description: Independent review facility PFS (IRF-PFS) is defined as the time from randomization to the first documented disease progression as determined by blinded independent central review with use of RECIST v1.1, or death due to any cause, whichever occurs first.
Time Frame: Randomization to first documented disease progression or death from any cause (up to 35 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin
Number analyzed (Participants) | 400 | 451
Months | 6.34 [6.24 to 8.05] | 7.10 [6.31 to 8.25]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab+Gemcitabine+Carboplatin/Cisplatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0373, Regression, Cox — inverse normal combination; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.73 to 1.01]

9. Secondary Outcome: OS Event Free Rate Atezolizumab+Gemcitabine+Carboplatin/Cisplatin Arm Versus Placebo+Gemcitabine+Carboplatin/Cisplatin Arm
Description: Overall Survival (OS) Event Free Rate at 1 Year.
Time Frame: Year 1
Population: The ITT population was defined as all participants randomized to the Atezolizumab+Gemcitabine+Carboplatin/Cisplatin or the Placebo+Gemcitabine+Carboplatin/Cisplatin arm in Stages 1 and 2, whether or not the assigned study treatment was received.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin
Number analyzed (Participants) | 400 | 451
Percentage | 55.00 [49.98 to 60.02] | 60.00 [55.39 to 64.61]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab+Gemcitabine+Carboplatin/Cisplatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1509, Z-test; Difference in Event Free Rate = 5.00, 95% CI 2-sided [-1.82 to 11.81]

10. Secondary Outcome: OS Event Free Rate in Atezolizumab Monotherapy Arm Versus Placebo+Gemcitabine+Carboplatin/Cisplatin Arm
Description: Overall Survival (OS) Event Free Rate at 1 Year.
Time Frame: Year 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 359 | 360
Percentage | 54.56 [49.23 to 59.88] | 57.91 [52.72 to 63.10]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab Monotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3761, Z-test; Difference in Event Free Rate = 3.36, 95% CI 2-sided [-4.08 to 10.79]

11. Secondary Outcome: PFS Event Free Rate
Description: Progression Free Survival (PFS) Event Free Rate at Year 1
Time Frame: Year 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin
Number analyzed (Participants) | 400 | 451
Percentage | 22.17 [17.93 to 26.42] | 30.47 [26.00 to 34.93]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab+Gemcitabine+Carboplatin/Cisplatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0083, Z-test; Difference in Event Free Rate = -8.29, 95% CI 2-sided [-14.45 to -2.13]

12. Secondary Outcome: Time to Deterioration in Global Health Status as Measured by the EORTC QLQ-C30 Score in the Placebo+Gemcitabine+Carboplatin/Cisplatin Arm Versus Atezolizumab +Gemcitabine+Carboplatin/Cisplatin Arm
Description: Time to deterioration in global health status as measured by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 in the Placebo+Gemcitabine+Carboplatin/Cisplatin Arm versus Atezolizumab +Gemcitabine+Carboplatin/Cisplatin Arm.
Time Frame: Up to approximately 73 months
Population: The patient reported outcome (PRO)-evaluable population is defined as participants in the ITT populations for comparisons of the Placebo+Chemo Arm versus Atezolizumab+Chemo Arm who have a baseline and at least one post-baseline assessment. The ITT population for the comparison of Atezo+Chemo Arm vs. Placebo+Chemo Arm included participants enrolled in Stage 1 and Stage 2, which consisted of 451 paarticipants in the Atezo+Chemo Arm and 400 participants in the Placebo+Chemo Arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin
Number analyzed (Participants) | 400 | 451
Months | 12.06 [8.28 to 20.24] | 32.07 [18.40 to NA] — Not evaluable due to sample size is very small and not enough events at later times to estimate the upper bound of the CI.
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab+Gemcitabine+Carboplatin/Cisplatin; Strata are: Enrollment Stage, PD-L1 Status, BAJORIN Risk Factor Score and Stratum 4 for all participants; Test type: Superiority; p = 0.0542, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.64 to 1.00]

13. Secondary Outcome: Time to Deterioration in Global Health Status as Measured by the EORTC QLQ-C30 Score in the Placebo+Gemcitabine+Carboplatin/Cisplatin Arm Versus Atezolizumab Monotherapy Arm
Description: Time to deterioration in global health status as measured by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 in the Placebo+Chemo Arm versus Atezolizumab Monotherapy Arm.
Time Frame: Up to approximately 73 months
Population: Evaluable population defined as patients in ITT for comparisons of Placebo+Chemo vs. Atezo Mono who have a baseline and at least one post-baseline assessment. ITT for comparison of Atezo Mono vs. Placebo+Chemo consisted of 360 patients enrolled in Atezo Mono in Stage 2. Although a total of 400 patients were randomized to Placebo+Chemo throughout study, only 359 patients who were concurrently enrolled into this arm in Stage 2 and prior to Protocol v6 were included in Placebo+Chemo of this ITT.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 359 | 360
Months | 12.02 [8.08 to 20.24] | 23.20 [8.31 to NA] — Not evaluable due to sample size is very small and not enough events at later times to estimate the upper bound of the CI.
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab Monotherapy; Strata are: PD-L1 Status, BAJORIN Risk Factor Score and Stratum 4 for all participants; Test type: Superiority; p = 0.6139, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.74 to 1.19]

14. Secondary Outcome: Time to Deterioration in Physical Function as Measured by the EORTC QLQ-C30 Score in the Placebo+Gemcitabine+Carboplatin/Cisplatin Arm Versus Atezolizumab +Gemcitabine+Carboplatin/Cisplatin Arm
Description: Median time to deterioration in physical function as measured by the QLQ-C30 in the Placebo+Gemcitabine+Carboplatin/Cisplatin Arm versus Atezolizumab +Gemcitabine+Carboplatin/Cisplatin Arm.
Time Frame: Up to approximately 73 months
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin
Number analyzed (Participants) | 400 | 451
Months | 15.74 [8.28 to 22.57] | 16.39 [9.07 to 26.68]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab+Gemcitabine+Carboplatin/Cisplatin; Strata are: Enrollment Stage, PD-L1 Status, BAJORIN Risk Factor Score and Stratum 4 for all participants; Test type: Superiority; p = 0.5540, Log Rank; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.86 to 1.32]

15. Secondary Outcome: Time to Deterioration in Physical Function as Measured by the EORTC QLQ-C30 Score in the Placebo+Gemcitabine+Carboplatin/Cisplatin Arm Versus Atezolizumab Monotherapy Arm
Description: Median time to deterioration in physical function as measured by the QLQ-C30 in the Placebo+Gemcitabine+Carboplatin/Cisplatin Arm versus Atezolizumab Monotherapy Arm.
Time Frame: Up to approximately 73 months
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 359 | 360
Months | 16.10 [8.08 to 22.57] | 9.23 [6.24 to 17.48]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab Monotherapy; Strata are: Enrollment Stage, PD-L1 Status, BAJORIN Risk Factor Score and Stratum 4 for all participants; Test type: Superiority; p = 0.0241, Log Rank; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [1.03 to 1.62]

16. Secondary Outcome: Maximum Atezolizumab Serum Concentration
Description: Maximum atezolizumab serum concentration.
Time Frame: Cycle 1 Day 1
Population: The pharmacokinetic (PK)-evaluable population is defined as all participants dosed with atezolizumab who have at least one post-baseline PK result.
Measure: Mean (Standard Deviation); unit: μg/ mL
Arm/Group | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 394 | 309
μg/ mL | 379 (125) | 390 (129)

17. Secondary Outcome: Minimum Atezolizumab Serum Concentration
Description: Minimum atezolizumab serum concentration.
Time Frame: Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 8 Day 1, Cycle 16 Day 1, Cycle 24 Day 1, Cycle 32 Day 1, Day 120 post dose of last blinded atezolizumab treatment, and study drug early discontinuation
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: μg/ mL
Arm/Group | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 382 | 297
μg/ mL
  Cycle 2 Day 1 | 79.8 (52.5) | 80.2 (46.0)
  Cycle 3 Day 1: number analyzed (Participants) | 365 | 245
  Cycle 3 Day 1 | 122 (47.2) | 129 (66.0)
  Cycle 4 Day 1: number analyzed (Participants) | 321 | 183
  Cycle 4 Day 1 | 153 (70.4) | 157 (63.4)
  Cycle 8 Day 1: number analyzed (Participants) | 194 | 104
  Cycle 8 Day 1 | 216 (96.8) | 193 (79.8)
  Cycle 16 Day 1: number analyzed (Participants) | 40 | 50
  Cycle 16 Day 1 | 235 (103) | 220 (79.8)
  Cycle 24 Day 1: number analyzed (Participants) | 36 | 29
  Cycle 24 Day 1 | 244 (75.7) | 233 (92.5)
  Cycle 32 Day 1: number analyzed (Participants) | 17 | 9
  Cycle 32 Day 1 | 259 (97.2) | 258 (60.5)
  Day 120 Post Dose of Last Blinded Atezo Trt: number analyzed (Participants) | 67 | 64
  Day 120 Post Dose of Last Blinded Atezo Trt | 18.8 (36.9) | 9.53 (12.7)
  Study Drug Early Discontinuation: number analyzed (Participants) | 194 | 148
  Study Drug Early Discontinuation | 154 (102) | 124 (83.8)

18. Secondary Outcome: Percentage of Participants With Anti-Therapeutic (Anti-Atezolizumab) Antibodies (ATAs)
Description: Percentage of participants with Anti-Therapeutic (Anti-Atezolizumab) Antibodies (ATAs).
Time Frame: Up to approximately 35 months
Population: The baseline ADA-evaluable population included participants who had a baseline ADA result. The post-baseline ADA-evaluable population included participants who had received at least one dose of the study treatment and who had at least one post-baseline ADA result.
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 434 | 341
Percentage of participants
  Baseline evaluable participants | 1.2 | 0.9
  Post-baseline evaluable participants: number analyzed (Participants) | 421 | 319
  Post-baseline evaluable participants | 19.7 | 26.3

19. Secondary Outcome: Investigator-Assessed Progression-Free Survival (INV-PFS) in Participants Treated With Atezolizumab Monotherapy Arm Compared With Placebo+Gemcitabine+Carboplatin/Cisplatin Arm
Description: as for outcome 1
Time Frame: Baseline up to disease progression, death, or loss of follow-up, whichever occurs first (assessed at baseline, every 9 weeks for 54 weeks and every 12 weeks thereafter up to 35 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 359 | 360
Months | 6.31 [6.24 to 6.74] | 2.69 [2.20 to 4.04]
Statistical Analysis 1: Comparison: Placebo+Gemcitabine+Carboplatin/Cisplatin vs Atezolizumab Monotherapy; Stratification factors: PD-L1 status and Bajorin risk score/presence of liver metastases and investigator choice of chemotherapy; Test type: Superiority; p = 1.0000, Log Rank; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [1.19 to 1.69]

20. Secondary Outcome: Percentage of Participants With Grade 3-4 Adverse Events (AEs)
Description: Percentage of participants with Grade 3-4 Adverse Events (AEs) assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Baseline up to 93 months
Population: The safety population was defined as participants who received any amount of any component of study treatment. Participants were analyzed according to the treatment received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 454 | 389 | 354
Percentage of Participants | 84.1 | 84.6 | 46.3

21. Secondary Outcome: Percentage of Participants With Grade 5 Adverse Events (AEs)
Description: Percentage of participants with Grade 5 Adverse Events (AEs) assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Baseline up to 93 months
Population: as for outcome 20
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 454 | 389 | 354
Percentage of Participants | 7.5 | 5.7 | 7.9

22. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: Percentage of participants with Serious Adverse Events (SAEs) assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Baseline up to 93 months
Population: as for outcome 20
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 454 | 389 | 354
Percentage of Participants | 53.7 | 50.6 | 46.0

23. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) Leading to Withdrawal of Any Study Treatment
Description: Percentage of participants with Adverse Events (AEs) leading to withdrawal of any study treatment assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Baseline up to 93 months
Population: as for outcome 20
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 454 | 389 | 354
Percentage of Participants | 36.3 | 33.9 | 9.0

24. Secondary Outcome: Percentage of Participants With Atezolizumab-Specific Adverse Events of Special Interest (AESIs)
Description: Percentage of participants with atezolizumab-specific Adverse Events of Special Interest (AESIs) Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Baseline up to 93 months
Population: as for outcome 20
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
Number analyzed (Participants) | 454 | 389 | 354
Percentage of Participants | 53.3 | 35.5 | 39.5

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 9 April 2024 (up to approximately 93 months)
Description: Serious & other adverse events reported based on safety population, which included patients who received any amount of any component of study treatment. There were 6 patients randomized to Atezo monotherapy after approval of Protocol version 6 who received open-label Atezo and chemo, and were pooled with patients in Atezo+chemo for safety analyses. All-cause mortality reported for deaths that occurred during study based on ITT, which included all randomized patients.
Arm/Group | Placebo+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin | Atezolizumab Monotherapy
All-Cause Mortality (participants affected / at risk) | 303/389 | 332/454 | 272/354
Serious Adverse Events (participants affected / at risk) | 197/389 | 244/454 | 163/354
Other Adverse Events (participants affected / at risk) | 379/389 | 441/454 | 300/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+Gemcitabine+Carboplatin/Cisplatin (N=389) | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin (N=454) | Atezolizumab Monotherapy (N=354)
Anaemia (Blood and lymphatic system disorders) | 19 (26) | 30 (34) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9) | 14 (15) | 0 (0)
Haematotoxicity (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Myelosuppression (Blood and lymphatic system disorders) | 3 (7) | 3 (6) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 8 (10) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4) | 6 (6) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (28) | 21 (30) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 3 (3) | 2 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (3)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 3 (3) | 7 (8)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (6) | 0 (0)
Accidental death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 4 (4) | 3 (3)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 7 (7) | 6 (6) | 2 (2)
Fatigue (General disorders) | 4 (4) | 3 (3) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 5 (6) | 4 (4)
Pyrexia (General disorders) | 12 (13) | 18 (19) | 9 (11)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Emphysematous pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Norovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 21 (24) | 8 (8)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 3 (3) | 1 (1) | 3 (3)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 4 (9) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Sepsis (Infections and infestations) | 8 (9) | 8 (9) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 30 (42) | 41 (62) | 22 (23)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 4 (4) | 3 (3) | 5 (5)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Stoma prolapse (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Urostomy complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 6 (7) | 4 (5) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 7 (8) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 12 (18) | 14 (23) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 3 (4) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Central nervous system haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Demyelination (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hemianopia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Miller Fisher syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 12 (12) | 15 (16) | 8 (8)
Anuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 10 (11) | 10 (11) | 13 (13)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 1 (1) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 3 (3) | 8 (8)
Renal impairment (Renal and urinary disorders) | 1 (1) | 5 (5) | 2 (2)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal tubular injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 3 (5) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary fistula (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 5 (5) | 4 (5)
Urinary tract obstruction (Renal and urinary disorders) | 3 (3) | 7 (7) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (9) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7) | 4 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (8) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Euthanasia (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Nephrostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Nephrostomy tube removal (Surgical and medical procedures) | 2 (2) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Leriche syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+Gemcitabine+Carboplatin/Cisplatin (N=389) | Atezolizumab+Gemcitabine+Carboplatin/Cisplatin (N=454) | Atezolizumab Monotherapy (N=354)
Anaemia (Blood and lymphatic system disorders) | 257 (481) | 308 (495) | 68 (83)
Leukopenia (Blood and lymphatic system disorders) | 64 (192) | 64 (132) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 148 (421) | 215 (510) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 117 (297) | 183 (378) | 12 (13)
Hyperthyroidism (Endocrine disorders) | 6 (6) | 35 (40) | 18 (20)
Hypothyroidism (Endocrine disorders) | 12 (12) | 44 (47) | 30 (31)
Abdominal pain (Gastrointestinal disorders) | 37 (54) | 43 (53) | 22 (27)
Constipation (Gastrointestinal disorders) | 111 (149) | 140 (187) | 67 (74)
Diarrhoea (Gastrointestinal disorders) | 73 (96) | 96 (146) | 42 (59)
Dyspepsia (Gastrointestinal disorders) | 22 (28) | 20 (21) | 5 (10)
Nausea (Gastrointestinal disorders) | 181 (317) | 202 (329) | 43 (53)
Vomiting (Gastrointestinal disorders) | 106 (175) | 122 (178) | 33 (43)
Asthenia (General disorders) | 98 (158) | 134 (208) | 51 (78)
Fatigue (General disorders) | 122 (182) | 134 (185) | 64 (83)
Malaise (General disorders) | 24 (35) | 18 (34) | 6 (6)
Oedema peripheral (General disorders) | 56 (68) | 53 (68) | 41 (56)
Pyrexia (General disorders) | 68 (113) | 122 (173) | 43 (57)
Nasopharyngitis (Infections and infestations) | 20 (25) | 33 (44) | 19 (31)
Upper respiratory tract infection (Infections and infestations) | 19 (26) | 30 (36) | 18 (22)
Urinary tract infection (Infections and infestations) | 61 (91) | 92 (141) | 59 (102)
Alanine aminotransferase increased (Investigations) | 26 (32) | 47 (58) | 24 (28)
Aspartate aminotransferase increased (Investigations) | 17 (28) | 48 (63) | 22 (26)
Blood alkaline phosphatase increased (Investigations) | 10 (15) | 27 (34) | 22 (29)
Blood creatinine increased (Investigations) | 45 (64) | 66 (89) | 28 (35)
Neutrophil count decreased (Investigations) | 129 (344) | 119 (331) | 0 (0)
Platelet count decreased (Investigations) | 138 (331) | 132 (350) | 5 (7)
Weight decreased (Investigations) | 25 (25) | 30 (35) | 23 (23)
White blood cell count decreased (Investigations) | 59 (165) | 62 (144) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 119 (165) | 144 (215) | 69 (72)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (21) | 26 (30) | 14 (35)
Hyperkalaemia (Metabolism and nutrition disorders) | 29 (39) | 24 (39) | 13 (19)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15 (24) | 21 (27) | 19 (20)
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 (27) | 26 (31) | 8 (16)
Hyponatraemia (Metabolism and nutrition disorders) | 16 (21) | 30 (36) | 9 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 (57) | 59 (84) | 42 (62)
Back pain (Musculoskeletal and connective tissue disorders) | 46 (57) | 56 (67) | 34 (40)
Myalgia (Musculoskeletal and connective tissue disorders) | 23 (34) | 27 (29) | 23 (30)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 (37) | 35 (43) | 22 (25)
Dizziness (Nervous system disorders) | 39 (51) | 45 (60) | 19 (20)
Headache (Nervous system disorders) | 34 (43) | 42 (65) | 25 (36)
Neuropathy peripheral (Nervous system disorders) | 23 (25) | 17 (19) | 6 (8)
Insomnia (Psychiatric disorders) | 34 (37) | 36 (39) | 19 (20)
Dysuria (Renal and urinary disorders) | 20 (26) | 29 (41) | 20 (23)
Haematuria (Renal and urinary disorders) | 51 (65) | 73 (104) | 48 (56)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (46) | 58 (67) | 30 (49)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 (43) | 43 (54) | 25 (29)
Alopecia (Skin and subcutaneous tissue disorders) | 49 (50) | 33 (35) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 33 (38) | 84 (123) | 41 (66)
Rash (Skin and subcutaneous tissue disorders) | 43 (52) | 91 (117) | 27 (32)
Hypertension (Vascular disorders) | 32 (42) | 46 (66) | 21 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-12-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT02807636/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT02807636/SAP_001.pdf